CLINICAL TRIAL: NCT07343635
Title: The Efficacy and Safety of Anti-inflammation Treatment (Hirudoid Introduction Followed by Yellow Light Therapy) Combined With Tofacitinib and Doxycycline in Chinese Adult Patients With Mild to Moderate Erythematous Telangiectatic Rosacea: A Prospective Parallel Controlled Single-blind Cohort Study
Brief Title: The Efficacy and Safety of Anti-inflammation Treatment (Hirudoid Introduction Followed by Yellow Light Therapy) Combined With Tofacitinib and Doxycycline in Chinese Adult Patients With Mild to Moderate Erythematous Telangiectatic Rosacea
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY-2025-274
Record Dates: First submitted 2025-12-04; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Erythematotelangiectatic Rosacea
MeSH Terms: conditions — Rosacea | interventions — Doxycycline; Hydroxychloroquine; tofacitinib

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): Participants receive doxycycline combined with hydroxychloroquine.
  Interventions: Drug: Doxycycline; Drug: Hydroxychloroquine
- Tofacitinib group (Active Comparator): Participants receive doxycycline combined with tofacitinib.
  Interventions: Drug: Doxycycline; Drug: Tofacitinib
- Anti-inflammation Treatment and Tofacitinib group (Experimental): Participants receive doxycycline and tofacitinib combined with anti-inflammatory treatment.
  Interventions: Drug: Doxycycline; Drug: Tofacitinib; Device: Anti-inflammatory Treatment (Hirudoid Introduction Followed by Yellow Light Therapy)

INTERVENTIONS:
Drug: Doxycycline — Doxycycline 100 mg orally once daily
Drug: Hydroxychloroquine — Hydroxychloroquine 200 mg orally twice daily.
  Arms: Control group
Drug: Tofacitinib — Tofacitinib 5mg orally twice daily.
  Arms: Anti-inflammation Treatment and Tofacitinib group; Tofacitinib group
Device: Anti-inflammatory Treatment (Hirudoid Introduction Followed by Yellow Light Therapy) — Topical application of Hirudoid followed by yellow light therapy (wavelength 590 nm, duration 20 minutes per session, once weekly)
  Arms: Anti-inflammation Treatment and Tofacitinib group

SUMMARY:
The efficacy and safety of anti-inflammation treatment (Hirudoid introduction followed by yellow light therapy) combined with tofacitinib and doxycycline in Chinese adult patients with mild to moderate erythematous telangiectatic rosacea: A prospective parallel controlled single-blind cohort study

ELIGIBILITY:
Inclusion Criteria:

* The subjects are male or female, aged 18 to 70 years (inclusive); they voluntarily participate in this study and sign the informed consent form.
* They are diagnosed with erythematous telangiectatic rosacea, meeting the diagnostic criteria in the "Chinese Guidelines for the Diagnosis and Treatment of Rosacea (2021)".
* At screening and baseline, the IGA score is 2 (mild) or 3 (moderate).
* The subjects agree not to use any other rosacea treatment drugs (prescription or over-the-counter) during the study period.
* The subjects are willing to minimize external factors that may trigger rosacea (such as spicy food, alcoholic beverages, prolonged sun exposure, etc.).
* The subjects (including their partners) agree that they have no plans to conceive within 3 months after signing the informed consent form until the end of the last treatment and are willing to take effective contraceptive measures voluntarily.

Exclusion Criteria:

* Diagnosed as papulopustular, hypertrophic, ocular rosacea or other special types of rosacea
* Other facial skin diseases that were active during the screening period or baseline may interfere with the efficacy/safety assessment of erythematous vasodilating rosacea, including but not limited to perioral dermatitis, facial keratosis, seborrheic dermatitis, and acne vulgaris. If the above-mentioned skin diseases were in clinical remission both during the screening period and at baseline, and the investigators determined that they would not affect the assessment of this study, they could be included.
* Subjects who have underlying known diseases or medical conditions, or who have undergone major surgeries within the six months prior to screening, where, based on the researcher's judgment, the subjects are at risk (such as cancer, leukemia or cachexia in the blood system);
* During the screening period or at baseline, researchers evaluate abnormal laboratory test results with significant clinical significance;
* Those who have received LED light therapy for their faces in the past two weeks;
* Those who have received laser, intense pulsed light (IPL), fractional microneedle radiofrequency treatment, CO2 exfoliating fractional laser treatment, electrocoagulation, dermabrasion, chemical peels, or any facial procedures (such as Thermage, etc.) for facial treatment in the past 6 weeks;
* Facial active infections who are currently receiving or require systemic treatment (systemic antibiotics, antifungal, antiviral drugs) - including bacterial pustules, fungal folliculitis, herpeder-like skin lesions and massive proliferation of Demodex mites;
* Local/systemic treatment that did not complete an adequate elution period before baseline, including: Glucocorticoids (corticosteroids), calcineurin inhibitors (such as tacrolimus, pimecrolimus), Janus kinase inhibitors, epidermal growth factors (such as commercially available repair dressings containing recombinant human EGF), acne treatment drugs (such as azelaic acid, retinoids, benzoyl peroxide, traditional Chinese medicine/Chinese patent medicine treatment), Such as tanshinone, metronidazole tablets, etc.), immunomodulators, topical astringents/exfoliating products, antibiotics (such as macrolides, metronidazole), high-concentration vitamin A (10,000 units per day), anti-pruritus drugs (such as antihistamines), etc.
* Use drugs that cause acne-like rashes simultaneously (such as azathioprine, haloperidol, halogens, lithium, systemic corticosteroids, phenytoin sodium, phenobarbital, testosterone, anabolic steroids, isoniazid);
* Those who have used astringents/exfoliating products (cleansing or exfoliating products containing salicylic acid or alcohol) within the past 2 days or are planned to use them during the study period;
* The subject has a history of alcohol abuse (drinking more than 14 units) within the past 2 years or a history of drug abuse within the past 5 years;
* Individuals infected with human immunodeficiency virus (HIV), those in the active stage of hepatitis C virus (HCV) infection (positive for anti-HCV), or those in the active stage of hepatitis B virus (HBV) infection (HBV-DNA > 2000IU/mL or 104 copies /ml), or those with positive Treponema pallidum antibodies showing an active stage of infection;
* Female subjects who plan to become pregnant or breastfeed during the study period;
* Those who are sensitive to light or use photosensitive drugs;
* People who are allergic to Hirudoid, tofacitinib, doxycycline, hydroxychloroquine or their ingredients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Achievement of IGA treatment success at Week 12 | 0 week、12 week
  Achievement of IGA treatment success(IGA = 0 or 1, and the proportion of subjects with an improvement of ≥2 grades from baseline) at Week 12

SECONDARY OUTCOMES:
The proportion of subjects achieving successful IGA treatment | From baseline to weeks 4, 8, and 12
  The proportion of subjects achieving successful IGA treatment (IGA = 0 or 1, and the proportion of subjects with an improvement of ≥2 grades from baseline)
Dermatology Life Quality Index（DLQI） | Baseline, week 12
  Patient questionnaire, score is calculated between 0 (worst score possible) and 30 (best score possible)
Change in facial erythema severity assessed by VISIA imaging system | From baseline to weeks 4, 8, and 12
  Facial erythema severity will be quantitatively assessed using the VISIA imaging system. Standardized facial photographs will be obtained at each visit, and changes in erythema severity from baseline will be evaluated using VISIA-derived analysis.